CLINICAL TRIAL: NCT02873611
Title: Estimation of the Localization Accuracy of the Genicular Ablation Procedure Applied for Chronic Pain Suppression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TPM Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CL-001-F1
Record Dates: First submitted 2016-07-24; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI scanning and the genicular ablation (Experimental): patients undergoing both MRI scanning and the genicular ablation procedure. additional MRI testing of apprx. 0.5-1 hour
  Interventions: Device: MRI; Procedure: genicular ablation procedure

INTERVENTIONS:
Device: MRI — patients will undergo an additional MRI testing of apprx. 0.5-1 hour.
Procedure: genicular ablation procedure

SUMMARY:
Estimation of the localization accuracy of the genicular ablation procedure applied for chronic pain suppression

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Diagnosed with primary degenerative osteoarthritis.
* Complaining of knee pains
* Patients clinically eligible for genicular nerve ablation procedure non-electively based on physical examination
* Patient signed ICF

Exclusion Criteria:

* Co-morbidities: patient suffers from neuropathy, bony tumors, traumatic fractures and DM.
* Claustrophobic or failing cooperativity assessment of laying still during long MRI scans
* Pregnancy or pregnancy suspicion
* Enrolled in concurrent studies that may confound the results of this study
* Clinical condition that in the investigator's opinion would not allow the subject to complete the study, e.g., tremor, extreme obesity, mental disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Location and orientation of the relevant genicular nerves based on eye-balling inspection of MRI images by a radiologist | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Fridman, MD, Principal Investigator — Assuta MC

IPD SHARING:
Plan to Share IPD: Undecided